CLINICAL TRIAL: NCT01023243
Title: Novel Use of Natural Language Processing and Targeted Patient Education Information Regarding the Process for Completion of the Foot Examination in Primary Care
Brief Title: Natural Language Processing and Quality Assessment in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Steven Smith, PI, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 08-002255
Record Dates: First submitted 2008-12-09; First posted 2009-12-02 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
Keywords: foot exam; health services; practice improvement; quality; preventive services; Natural Language Processing
MeSH Terms: conditions — Diabetes Mellitus | interventions — Tobacco Products

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 CAre of the Feet for Those at Risk (Placebo Comparator): secular trends for physician documentation in the medical record for care of the feet for high risk patients
  Interventions: Other: Brochure: Care of the Feet for Those at Risk; Other: Quality Survey: foot exam, tobacco and aspirin use
- Care of the feet for those at risk (Active Comparator): the impact of 1) patient survey regarding last foot exam, tobacco and aspirin use on documentation of foot exam and 2) patient education material: Care of the Foot For Those at Risk, on documentation of foot examination in the medical record
  Interventions: Other: Quality Survey: foot exam, tobacco and aspirin use
- Impact of Quality Survey (Active Comparator): Impact of patient survey regarding last foot exam, tobacco and aspirin use on documentation of foot exam in the medical record
  Interventions: Other: Brochure: Care of the Feet for Those at Risk

INTERVENTIONS:
Other: Brochure: Care of the Feet for Those at Risk — Patient education materials and key messages for care of the feet for those patients at risk
  Other Names: Care of the Feet For Those at Risk
  Arms: 1 CAre of the Feet for Those at Risk; Impact of Quality Survey
Other: Quality Survey: foot exam, tobacco and aspirin use — NCQA Patient Survey
  Other Names: Care of the Feet For Those at Risk
  Arms: 1 CAre of the Feet for Those at Risk; Care of the feet for those at risk

SUMMARY:
The investigators propose to use a Natural Language Processing System (NLP) to provide an initial baseline report for primary care patients at risk for diabetes and cardiovascular complications that will include: a) evidence of foot exam documentation in the previous year; b) use of aspirin for cardiovascular risk reduction; and c) tobacco use. As part of a randomized trial, we plan to use a previously validated mailed survey (NCQA Provider Recognition Program) that requests information on the last foot exam, use of aspirin and tobacco. Patients who have been identified by NLP as not having had a foot exam will be randomized into treatment and control arms. Both arms will receive an informational letter; with a second mailing to nonresponders after one month, describing the key strategies for effective patient-physician communication during the clinical encounter. The treatment arm will also receive an informational letter and patient education brochure containing key messages about the importance of regular foot examinations. NLP will be repeated after 6 months to compare the impact of the patient education materials.

ELIGIBILITY:
Inclusion Criteria:

* primary care patients with diagnosis of diabetes

Exclusion Criteria:

* unwilling to give informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Completion of foot exam | 6 months post intervention

SECONDARY OUTCOMES:
Patient report in validation of Natural Language Processing | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory a Bartel, MD, Principal Investigator — Mayo Clinic; Steven A Smith, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Pakhomov S, Bjornsen S, Hanson P, Smith S. Quality performance measurement using the text of electronic medical records. Med Decis Making. 2008 Jul-Aug;28(4):462-70. doi: 10.1177/0272989X08315253. Epub 2008 May 13. PMID 18480037